CLINICAL TRIAL: NCT03148002
Title: An Evaluation of the Efficacy and Safety of a Polyethylene Glycol (PEG) Based Bowel Protocol for the Management of Constipation in Peritoneal Dialysis Patients: A Pilot Study
Brief Title: Peritoneal Dialysis Pilot Study: Evaluating Polyethylene Glycol (PEG) for Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDBowel2017
Record Dates: First submitted 2017-03-14; First posted 2017-05-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Constipation; Peritoneal Dialysis Complication
MeSH Terms: conditions — Constipation | interventions — Sennosides; Lactulose; Phenolphthalein

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to received the Current Bowel Protocol or the PEG Bowel Protocol
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Current Bowel Protocol (Active Comparator): Patients will receive the Current Bowel Protocol with senna. Lactulose will be used for rescue therapy.
  Interventions: Drug: Current Bowel Protocol (senna/lactulose)
- PEG Bowel Protocol (Active Comparator): Patients will receive the Protocol with Polyethylene Glycol 3350. Lactulose will be used for rescue therapy.
  Interventions: Drug: PEG Bowel Protocol (PEG/lactulose)

INTERVENTIONS:
Drug: Current Bowel Protocol (senna/lactulose) — Stimulant and Osmotic Laxatives.
  Other Names: Senna; Lactulose; Sennosides; DIN 02242814; DIN: 02412268; NPN: 00367729; NPN: 00026158
  Arms: Current Bowel Protocol
Drug: PEG Bowel Protocol (PEG/lactulose) — Osmotic Laxatives.
  Other Names: PEG; Lax-A-Day; Pegalax; DIN: 02328232; Restoralax; DIN: 02318164; DIN: 02317680; Lactulose; DIN 02242814; DIN: 02412268
  Arms: PEG Bowel Protocol

SUMMARY:
Constipation is a common condition, which occurs one in four Canadians. Maintaining regular bowel movements is imperative because constipation can affect the quality of PD dialysate flow and result in an unwanted effect on the dialysis adequacy.

There is limited data on how to best manage constipation in the peritoneal dialysis population. Polyethylene glycol (PEG) is an osmotic laxative that is becoming popular for prevention and treatment of constipation across Canada. Although some PD programs in Canada have already converted to PEG for management of constipation, more research in this population would help guide practice. For now, the current PD bowel regimen at the Nova Scotia Health Authority (NSHA) includes daily preventative therapy using a stimulant laxative, senna, along with an osmotic laxative, lactulose, for acute constipation.

The investigators will review all patients in the NSHA PD program who have regular or recent laxative use for participation in this study. Patients included in this study will be randomly assigned to the Current Bowel Protocol or the PEG Bowel Protocol for 8 weeks.

The goal is to determine if the PEG Bowel Protocol is as effective and safe for the prevention of constipation as the Current Bowel Protocol used in the PD Program. The investigators will use bowel function diaries and patient surveys to determine efficacy and safety outcomes.

DETAILED DESCRIPTION:
Constipation is a common condition, which impacts one in four Canadians Maintaining regular bowel movements is important in the peritoneal dialysis (PD) population because constipation can negatively impact the quality of dialysate flow and can result in impaired dialysis adequacy. Unfortunately, treating constipation is challenging in PD patients because of the diet and fluid restrictions required in this population, as well as the need for constipating calcium based phosphate binders.

Constipation treatment can be administered orally or rectally. Although patients often prefer oral therapy, there are occasions when rectal therapy is preferred (ie. rectal suppositories and enemas). Oral laxatives include bulk, osmotic, stimulant, and lubricants.

In the Nova Scotia (NS) PD Program, patients are counseled to maintain a type 3-4 stool on the Bristol Stool Chart (BSC). An ideal stool is a type 4, which appears like a sausage or snake and is smooth and soft in consistency. To maintain a type 3-4 stool, current therapy includes senna 8.6-17.2 g twice daily with the addition of lactulose 30-60 mL twice daily, as needed. Rescue therapy in the Current Bowel Protocol is lactulose 30-60 mL every hour until bowel movement.

There is limited evidence to guide the ideal bowel regimen in PD patients. Reasons to consider PEG therapy include the evidence promoting PEG in the general population with constipation, the positive outcomes found in a small population of PD patients (Mimidis 2005), as well as positive feedback from other provinces who currently recommend PEG in PD patients. The investigators postulate the PEG protocol would be as effective and safe as the Current Bowel Protocol, and thus will evaluate PEG in the PD population, the investigators will conduct a prospective, interventional, randomized, open label, pilot study.

All patients with recent laxative use will be approached for inclusion. Patients will be randomly assigned to the Current Bowel Protocol (senna/lactulose) or the PEG Bowel Protocol (PEG/lactulose) for 8 weeks.

The primary objective is to compare the efficacy of the PEG Bowel Protocol in preventing constipation to the Current Bowel Protocol. We will review the safety of the regimens by monitoring for adverse events from all laxatives and explore the impact of constipation in patients who experience PD treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the peritoneal dialysis program in Nova Scotia who are currently taking laxatives.

Exclusion Criteria:

* Allergy or intolerance to any of the study laxatives (PEG, senna, lactulose); cognitive impairment or inability to document symptoms; known or suspected gastrointestinal obstruction or ileus; known or planned pregnancy; no laxative use in the last 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Rate of constipation treatment success | 8 weeks.
  Successful treatment of constipation will be defined based on a modified ROME criteria developed by Dipalma 2007: relief of constipation for more than 50% of the weeks in the study.

SECONDARY OUTCOMES:
Number of patients with laxative related adverse effects. | 8 weeks.
  Compare the occurrence of side effects during the study period.
Mean change from baseline on the PAC-SYM questionnaire | 8 weeks.
  Measure of the impact of constipation disease severity. PAC-SYM = Patient Assessment of Constipation Symptoms (Frank 1999 and Bove 2012)
Mean change from baseline on the PAC-QOL questionnaire | 8 weeks
  Measure the impact of constipation on quality of life. PAC-QOL = Patient Assessment of Constipation Quality of Life (Marquis 2005 and Bove 2012)
Incidence of peritoneal dialysis treatment failure requiring intervention | 8 weeks
  Interventions include antibiotics for peritonitis, catheter re-positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Y Tran, BScPharm, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mimidis K, Mourvati E, Kaliontzidou M, Papadopoulos V, Thodis E, Kartalis G, Vargemezis V. Efficacy of polyethylene glycol in constipated CAPD patients. Perit Dial Int. 2005 Nov-Dec;25(6):601-3. No abstract available. PMID 16411529
- [Background] Setyapranata S, Holt SG. The Gut in Older Patients on Peritoneal Dialysis. Perit Dial Int. 2015 Nov;35(6):650-4. doi: 10.3747/pdi.2014.00341. PMID 26702007
- [Background] Pare P, Ferrazzi S, Thompson WG, Irvine EJ, Rance L. An epidemiological survey of constipation in canada: definitions, rates, demographics, and predictors of health care seeking. Am J Gastroenterol. 2001 Nov;96(11):3130-7. doi: 10.1111/j.1572-0241.2001.05259.x. PMID 11721760
- [Background] Sutton D, Dumbleton S, Allaway C. Can increased dietary fibre reduce laxative requirement in peritoneal dialysis patients? J Ren Care. 2007 Oct-Dec;33(4):174-8. doi: 10.1111/j.1755-6686.2007.tb00068.x. PMID 18298035
- [Background] Sutton D, Ovington S, Engel B. A multi-centre, randomised trial to assess whether increased dietary fibre intake (using a fibre supplement or high-fibre foods) produces healthy bowel performance and reduces laxative requirement in free living patients on peritoneal dialysis. J Ren Care. 2014 Sep;40(3):157-63. doi: 10.1111/jorc.12056. Epub 2014 Mar 20. PMID 24650128
- [Background] Dessau RB, Olsen OB, Frifelt JJ, Skott H. Influence of psyllium seed husk on azotemia, electrolytes, and bowel regulation in patients on CAPD. Perit Dial Int. 1989;9(4):351. No abstract available. PMID 2488394
- [Background] Pare P. The approach to diagnosis and treatment of chronic constipation: suggestions for a general practitioner. Can J Gastroenterol. 2011 Oct;25 Suppl B(Suppl B):36B-40B. doi: 10.1155/2011/368189. PMID 22114756
- [Background] Liu LW. Chronic constipation: current treatment options. Can J Gastroenterol. 2011 Oct;25 Suppl B(Suppl B):22B-28B. PMID 22114754
- [Background] Schuster BG, Kosar L, Kamrul R. Constipation in older adults: stepwise approach to keep things moving. Can Fam Physician. 2015 Feb;61(2):152-8. No abstract available. PMID 25676646
- [Background] Ramkumar D, Rao SS. Efficacy and safety of traditional medical therapies for chronic constipation: systematic review. Am J Gastroenterol. 2005 Apr;100(4):936-71. doi: 10.1111/j.1572-0241.2005.40925.x. PMID 15784043
- [Background] Hsieh C. Treatment of constipation in older adults. Am Fam Physician. 2005 Dec 1;72(11):2277-84. PMID 16342852
- [Background] Di Palma JA, Smith JR, Cleveland Mv. Overnight efficacy of polyethylene glycol laxative. Am J Gastroenterol. 2002 Jul;97(7):1776-9. doi: 10.1111/j.1572-0241.2002.05840.x. PMID 12135034
- [Background] Attar A, Lemann M, Ferguson A, Halphen M, Boutron MC, Flourie B, Alix E, Salmeron M, Guillemot F, Chaussade S, Menard AM, Moreau J, Naudin G, Barthet M. Comparison of a low dose polyethylene glycol electrolyte solution with lactulose for treatment of chronic constipation. Gut. 1999 Feb;44(2):226-30. doi: 10.1136/gut.44.2.226. PMID 9895382
- [Background] Lee-Robichaud H, Thomas K, Morgan J, Nelson RL. Lactulose versus Polyethylene Glycol for Chronic Constipation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007570. doi: 10.1002/14651858.CD007570.pub2. PMID 20614462
- [Background] Christie AH, Culbert P, Guest JF. Economic impact of low dose polyethylene glycol 3350 plus electrolytes compared with lactulose in the management of idiopathic constipation in the UK. Pharmacoeconomics. 2002;20(1):49-60. doi: 10.2165/00019053-200220010-00005. PMID 11817992
- [Background] Taylor RR, Guest JF. The cost-effectiveness of macrogol 3350 compared to lactulose in the treatment of adults suffering from chronic constipation in the UK. Aliment Pharmacol Ther. 2010 Jan 15;31(2):302-12. doi: 10.1111/j.1365-2036.2009.04191.x. Epub 2009 Nov 3. PMID 19886948
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Bove A, Pucciani F, Bellini M, Battaglia E, Bocchini R, Altomare DF, Dodi G, Sciaudone G, Falletto E, Piloni V, Gambaccini D, Bove V. Consensus statement AIGO/SICCR: diagnosis and treatment of chronic constipation and obstructed defecation (part I: diagnosis). World J Gastroenterol. 2012 Apr 14;18(14):1555-64. doi: 10.3748/wjg.v18.i14.1555. PMID 22529683
- [Background] Yiannakou Y, Piessevaux H, Bouchoucha M, Schiefke I, Filip R, Gabalec L, Dina I, Stephenson D, Kerstens R, Etherson K, Levine A. A randomized, double-blind, placebo-controlled, phase 3 trial to evaluate the efficacy, safety, and tolerability of prucalopride in men with chronic constipation. Am J Gastroenterol. 2015 May;110(5):741-8. doi: 10.1038/ajg.2015.115. Epub 2015 Apr 14. PMID 25869393
- [Background] Dipalma JA, Cleveland MV, McGowan J, Herrera JL. A randomized, multicenter, placebo-controlled trial of polyethylene glycol laxative for chronic treatment of chronic constipation. Am J Gastroenterol. 2007 Jul;102(7):1436-41. doi: 10.1111/j.1572-0241.2007.01199.x. Epub 2007 Mar 31. PMID 17403074
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Gokal R, Alexander S, Ash S, Chen TW, Danielson A, Holmes C, Joffe P, Moncrief J, Nichols K, Piraino B, Prowant B, Slingeneyer A, Stegmayr B, Twardowski Z, Vas S. Peritoneal catheters and exit-site practices toward optimum peritoneal access: 1998 update. (Official report from the International Society for Peritoneal Dialysis). Perit Dial Int. 1998 Jan-Feb;18(1):11-33. No abstract available. PMID 9527026